CLINICAL TRIAL: NCT02740907
Title: Premolar Autotransplantation in Juvenile Dentition: Quantitative Assessment of Vertical Bone and Soft Tissue Growth
Status: Completed | Type: Observational
Sponsor: MKG-Praxisklinik (Other)
Responsible Party: Principal Investigator, Dirk Nolte, MD DDS PhD, Dirk Nolte, MD DDS PhD, MKG-Praxisklinik
Other Study IDs: Premolar transplantation
Record Dates: First submitted 2016-03-22; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Traumatic Dental Injury; Tooth Aplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: premolar autotransplantation — Autogenous tooth transplantation of premolars to the anterior maxilla to stimulate bone and soft tissue growth.

SUMMARY:
Objective:

Premolar autotransplantation represents an effective therapeutic option for the treatment of juvenile dentition in traumatic dental injury with tooth loss. Numerous studies report on the osteoinductive potency of the method, however, to date no quantitative data has been provided. The objective of this prospective clinical study was to quantitatively assess the bone and soft tissue levels after autogenous premolar transplantation by clinical and radiographic parameters.

Materials/Methods:

In the study 26 premolars were transplanted in 20 patients after traumatic dental injury (n=10) or tooth aplasia (n=16) in the upper front. Standard clinical parameters were evaluated. Based on a standardized photo documentation, the relative soft tissue level was measured in comparison to the healthy adjacent teeth. Radiographic findings involved the evaluation of root resorption, pulp canal obliterations and the relative bone height. Patient satisfaction was determined using a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* premolar transplantation after tooth loss in the anterior maxilla (13-23) by aplasia or trauma

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients (mean age 13.6, f:10, m:10) suffering from tooth loss in the anterior maxilla (13-23). Thirteen patients suffered from traumatic dental injury (TDI) with subsequent tooth loss (n=16 transplants). In 7 patients, aplasia of teeth in region 13 to 23 was present (n=10 transplants).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Transplant survival | 2006-2014
  Evaluation by Kaplan-Meier-Estimator.
Soft tissue development | 2006-2014
  Measurement by standardized clinical documentation.
Bone development | 2006-2014
  Measurement by radiographic evaluation.
Sensibility | 2006-2014
  Assessment of clinical sensibility.
Root resorptions | 2006-2014
  Radiographic evaluation.
Pulp obliteration | 2006-2014
  Radiographic evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- MKG Praxisklinik, Munich, Sauerbruchstraße 48, Germany

IPD SHARING:
Plan to Share IPD: No